CLINICAL TRIAL: NCT00932971
Title: A Multicenter Randomised Study Comparing the Efficacy of PegIFN-alfa2a Plus Placebo vs. PegIFN-alfa2a Plus Tenofovir for the Treatment of Chronic Delta Hepatitis-The Hep-Net International Delta Hepatitis Interventional Trial II (HIDIT-II)
Brief Title: HIDIT II - PegIFN-alfa2a Plus Tenofovir in Chronic Delta Hepatitis
Acronym: HIDIT-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HepNet Study House, German Liverfoundation (Network)
Collaborators: Hannover Medical School (Other); Hoffmann-La Roche (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hep-Net-HIDIT-II; EudraCT-No.: 2008-005560-13
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — peginterferon alfa-2a; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-IFN alfa-2a plus placebo (Placebo Comparator): Pegylated interferon alfa-2a 180 µg once weekly (QW) subcutaneous (sc) plus placebo once daily, orally
  Interventions: Drug: PEG-IFN alfa-2a, placebo
- PEG-IFN alfa-2a plus Tenofovir (Active Comparator): Pegylated interferon alfa-2a 180 µg once weekly (QW) subcutaneous (sc) plus Tenofovir disoproxilfumarat 245mg once daily, orally
  Interventions: Drug: PEG-IFN alfa-2a, Tenofovir

INTERVENTIONS:
Drug: PEG-IFN alfa-2a, Tenofovir — Pegylated interferon alfa-2a, 180µg once weekly, subcutaneously; Tenofovir disoproxilfumarat, 245mg, once daily, orally
  Other Names: Pegasys; Viread
  Arms: PEG-IFN alfa-2a plus Tenofovir
Drug: PEG-IFN alfa-2a, placebo — Pegylated interferon alfa-2a, 180µg once weekly, subcutaneously; Placebo, once daily, orally
  Other Names: Pegasys
  Arms: PEG-IFN alfa-2a plus placebo

SUMMARY:
Randomized, double blind study comparing the efficacy of pegylated interferon-alfa2a plus placebo versus pegylated interferon-alfa2a plus tenofovir for the treatment of chronic delta hepatitis. 70 Patients will be randomized 1:1 into the two groups. Treatment duration: 96 weeks. Follow-up: 24 weeks. Long-term-follow-up: until week 358.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age > 18 years.
* Positive HBsAg, for at least the prior 6 months, positive anti-HDV for at least 3 months and positive for HDV-RNA by PCR within the screening period.
* Elevated serum ALT ≥ ULN but ≤ 10X ULN as determined by two abnormal values taken > 1 month apart during the 12 months before the first dose of study drug with at least one of the determinations obtained ≤ 35 days prior to the first dose.
* A liver biopsy obtained within the past 12 months demonstrating liver disease consistent with chronic hepatitis. Patients with cirrhosis on liver biopsy must also have a liver imaging investigation to rule out hepatic carcinoma.
* Negative urine or serum pregnancy test documented within the 24 hour period prior to the first dose of test drug.
* Additionally, all fertile males with partners of childbearing age and females should use two reliable forms of effective contraception (combined) throughout the entire period of the study (treatment and for 4 months after treatment completion)
* Creatinine clearance ≥ 70 mL/min

Exclusion Criteria:

* Patients must not have received antiviral therapy for their chronic hepatitis D within the previous 6 months. Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study are also excluded.
* Positive test at screening for HAV-Ag-IgM, HCV-RNA or HCV-Ag or HIV-Ag.
* Serum concentrations of ceruloplasmin or alpha-1-antitrypsin consistent with an increased risk of metabolic liver disease.
* Evidence of decompensated liver disease (Childs B-C).
* History or other evidence of a medical condition associated with chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures, thalassemia).
* Women with ongoing pregnancy or who are breast feeding.
* WBC count of < 3.000 cells/ mm3; neutrophil count < 1.500 cells/mm3or platelet count < 90.000 cells/mm3.
* Evidence of alcohol and/or drug abuse within one year of entry.
* Patients are excluded if any history of psychiatric disease, especially depression, or of suicidal attempts is evident.
* History of immunologically mediated disease.
* History or other evidence of decompensated liver disease.
* History or other evidence of chronic pulmonary disease associated with functional limitation.
* History of severe cardiac disease
* Evidence of an active or suspected cancer or a history of malignancy where there is a risk of cancer to recur.
* History of having received any systemic anti-neoplastic (including radiation) or immunomodulatory treatment (including systemic corticosteroids) ≤ 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* History of any organ transplantation with an existing functional graft
* History of thyroid disease poorly controlled on prescribed medications. Patients with elevated thyroid stimulating hormone concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded.
* History or evidence of severe retinopathy or clinically relevant ophthalmological disorder.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* Patients with a value of alpha-fetoprotein >100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months.
* History or evidence for any intolerance or hypersensitivity to pegylated interferon-alfa-2a, tenofovir or other substances part of the study medication.
* Current participation in any other investigational trial and participation in another investigational trial within 3 months before the trial begins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Negativation of HDV-RNA at the end of therapy | week 96

SECONDARY OUTCOMES:
Negativation of HDV-RNA at week 48 of treatment | week 48
Negativation of HDV-RNA 24 weeks after the end of treatment | week 120
Normalization of ALT levels at the end of treatment and at the end of follow-up | week 96 and week 356
HDV-RNA-levels over time | up to week 356
Suppression of HBV-DNA below 6 IU/ml using the Cobas TaqMan assay at treatment weeks 48 and 96 and 24 weeks after treatment | week 48, week 96, week 120
Liver histology at end of treatment (Ishak score for inflammation and fibrosis) | week 96
Quantitative HBsAg levels over time. Loss of HBsAg and development of anti-HBs antibodies, intrahepatic cccDNA and HBV-DNA levels over time | up to week 356
HBV- and HDV-virus-specific T cell responses during therapy and after 24 weeks of follow up if virological and biochemical efficacy has been shown | up week 120
Virological long-term outcome | 1, 2, 3, 4 and 5 years after the end of treatment
Clinical long-term outcome | 1, 2, 3, 4 and 5 years after the end of treatment
Quality of Life | up to week 356

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Manns, Prof. Dr., Study Director — Hannover Medical School
Locations (10):
- Germany (7):
  - Charité Campus Virchow-Klinikum, Med. Klinik für Gastroenterologie und Hepatologie, Berlin
  - Friedrich-Wilhelms-Universität, Med. Klinik und Poliklinik I, Bonn
  - Universitätsklinikum Düsseldorf, Klinik für Gastroenterologie, Düsseldorf
  - Klinikum der J.W. Goethe-Universität, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Innere Medizin, Hamburg
  - Medizinische Hochschule Hannover, Zentrum Innere Medizin, Hanover
  - Medizinische Fakultät der Universität Heidelberg, Innere Medizin IV, Heidelberg
- Athens University School of Medicine, Hippokration General Hospital, Athens, Greece
- Romania (2):
  - Institutul de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Spitalul Clinic de Boli Infectioase si, Timișoara

REFERENCES:
- [Background] Heidrich B, Deterding K, Tillmann HL, Raupach R, Manns MP, Wedemeyer H. Virological and clinical characteristics of delta hepatitis in Central Europe. J Viral Hepat. 2009 Dec;16(12):883-94. doi: 10.1111/j.1365-2893.2009.01144.x. Epub 2009 Jun 28. PMID 19566789
- [Background] Wedemeyer H, Yurdaydin C, Dalekos GN, Erhardt A, Cakaloglu Y, Degertekin H, Gurel S, Zeuzem S, Zachou K, Bozkaya H, Koch A, Bock T, Dienes HP, Manns MP; HIDIT Study Group. Peginterferon plus adefovir versus either drug alone for hepatitis delta. N Engl J Med. 2011 Jan 27;364(4):322-31. doi: 10.1056/NEJMoa0912696. PMID 21268724
- [Background] Heidrich B, Yurdaydin C, Kabacam G, Ratsch BA, Zachou K, Bremer B, Dalekos GN, Erhardt A, Tabak F, Yalcin K, Gurel S, Zeuzem S, Cornberg M, Bock CT, Manns MP, Wedemeyer H; HIDIT-1 Study Group. Late HDV RNA relapse after peginterferon alpha-based therapy of chronic hepatitis delta. Hepatology. 2014 Jul;60(1):87-97. doi: 10.1002/hep.27102. PMID 24585488
- [Derived] Yurdaydin C, Kahlhofer J, Caruntu FA, Yalcin K, Gurel S, Akarca US, Sprinzl K, Bock HH, Bockmann JH, Papatheodoridis GV, Merle U, Demir M, Hardtke S, Keskin O, Idilman R, Cornberg M, Wedemeyer H, Wranke A. Ten-Year Follow-Up After 96 Weeks Treatment With Peginterferon Plus Tenofovir in Hepatitis D (HIDIT-II): Improved Clinical Outcome After Combination Therapy. United European Gastroenterol J. 2026 Feb;14(1):e70153. doi: 10.1002/ueg2.70153. Epub 2025 Nov 29. PMID 41317314
- [Derived] Hardtke S, Yurdaydin C, Caruntu FA, Curescu MG, Yalcin K, Akarca US, Gurel S, Zeuzem S, Erhardt A, Luth S, Papatheodoridis GV, Port K, Manns MP, Cornberg M, Kahlhofer J, Wedemeyer H. Frequency, Severity and Impact of Pegylated Interferon Alpha-Associated Flares in Hepatitis D Infection. J Viral Hepat. 2025 Apr;32(4):e70022. doi: 10.1111/jvh.70022. PMID 40087915
- [Derived] Anastasiou OE, Caruntu FA, Curescu MG, Yalcin K, Akarca US, Gurel S, Zeuzem S, Erhardt A, Luth S, Papatheodoridis GV, Keskin O, Port K, Radu M, Celen MK, Idilman R, Heidrich B, Mederacke I, von der Leyen H, Kahlhofer J, von Karpowitz M, Hardtke S, Cornberg M, Yurdaydin C, Wedemeyer H. Five-year follow-up of 96 weeks peginterferon plus tenofovir disoproxil fumarate in hepatitis D. Liver Int. 2024 Jan;44(1):139-147. doi: 10.1111/liv.15745. Epub 2023 Oct 3. PMID 37787009
- [Derived] Wedemeyer H, Yurdaydin C, Hardtke S, Caruntu FA, Curescu MG, Yalcin K, Akarca US, Gurel S, Zeuzem S, Erhardt A, Luth S, Papatheodoridis GV, Keskin O, Port K, Radu M, Celen MK, Idilman R, Weber K, Stift J, Wittkop U, Heidrich B, Mederacke I, von der Leyen H, Dienes HP, Cornberg M, Koch A, Manns MP; HIDIT-II study team. Peginterferon alfa-2a plus tenofovir disoproxil fumarate for hepatitis D (HIDIT-II): a randomised, placebo controlled, phase 2 trial. Lancet Infect Dis. 2019 Mar;19(3):275-286. doi: 10.1016/S1473-3099(18)30663-7. PMID 30833068
- [Derived] Bremer B, Anastasiou OE, Ciesek S, Wedemeyer H. Automated nucleic acid isolation methods for HDV viral load quantification can lead to viral load underestimation. Antivir Ther. 2019;24(2):117-123. doi: 10.3851/IMP3281. PMID 30516520
- See also: Related Info — http://www.kompetenznetz-hepatitis.de
- See also: Related Info — http://www.hepatitis-delta.org